CLINICAL TRIAL: NCT00178477
Title: Feasibility Study for Gated External-Beam Radiotherapy for Patients With Internal, Extra-cranial Tumors
Brief Title: Study of Breath-holding as a Means to Reduce Tumor Motion From Breathing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Drs Okunieff and ODell have left the University of Rochester
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URCC 3701
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Neoplasm, Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Magnetic Resonance Spectroscopy; Breath Holding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breath-holding (Experimental): MRI with breath-holding
  Interventions: Procedure: MRI with breath-holding

INTERVENTIONS:
Procedure: MRI with breath-holding — Breath holding for diminished tumor motion.

SUMMARY:
The purpose of this research study is to evaluate typical tumor motion caused by breathing using MRI and can help determine whether simple passive breathing and/or breath-holding could be used for the future treatment of similar lung and liver tumors using radiation therapy radiosurgery techniques.

ELIGIBILITY:
Inclusion Criteria:

* The patient is enrolled on U8700 RSRB # A Phase II Study For Using Radiosurgery On Limited Metastases Of Breast Cancer or U9700 A Pilot Study For Using Radiosurgery On Limited Metastases.
* ≥ 18 years of age
* has given Informed consent

Exclusion Criteria:

-Contraindications for any MRI procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter O'Dell, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Department of Radiation Oncology, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be identified from patients seen in the Department of Radiation Oncology and who have previously consented to participate in URCC 8700 or URCC 9700.
Groups:
- Breath Hold: MRI with Breath Hold
Period: Overall Study
Arm/Group | Breath Hold
Started | 10
Completed | 5
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- Group 1: MRI with Breath Hold
Arm/Group | Group 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Tumor Motion Related to Breathing as Determined From MRI Images
Description: 1. Determine the typical and maximal tumor 3D displacements over the respiratory cycle and how these values vary depending on the tumor location
  2. Determine the reproducibility of target position over multiple breath-holds
  3. Determine the variability across patients in respiratory-derived lesion motion and target position reproducibility over multiple breath-holds
Time Frame: 20 - 30 seconds
Population: Data were not analyzed due to study termination.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No